CLINICAL TRIAL: NCT05446272
Title: The Diaphragmatic Initiated Ventilatory Assist (DIVA) Trial
Acronym: DIVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 849912
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Extubation Failure; Bronchopulmonary Dysplasia; Death
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Death

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Trial PIs are unaware of treatment allocation for individual subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NIV-NAVA (Experimental)
  Interventions: Device: NIV-NAVA
- NS- NIPPV (Active Comparator)
  Interventions: Device: NS-NIPPV

INTERVENTIONS:
Device: NIV-NAVA — Infants in the intervention arm will be managed with non-invasive neurally adjusted ventilatory assist (NIV-NAVA) using FDA-approved servos with associated FDA-approved Edi catheter.
  Other Names: Non-invasive Neurally Adjusted Ventilatory Assist
  Arms: NIV-NAVA
Device: NS-NIPPV — Infants in the active comparator arm will be treated with non-synchronized non-invasive positive pressure ventilation (NIPPV) through FDA-approved ventilators currently in use at each site.
  Other Names: Non-synchronized Non-invasive Positive Pressure Ventilation
  Arms: NS- NIPPV

SUMMARY:
DIVA is a pragmatic randomized clinical trial (RCT) to determine: among (P) preterm infants born 23 0/7-28 6/7 weeks gestation undergoing extubation from mechanical ventilation, whether (I) Non-invasive neurally adjusted ventilatory assist (NIV-NAVA) (C) compared with Non-synchronized nasal intermittent positive pressure ventilation (NS-NIPPV), will reduce the incidence of (O) extubation failure within (T) 5 days (120 hours) of extubation.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is the most common complication of prematurity and is the leading respiratory cause of childhood morbidity. Ventilator induced lung injury (VILI) an accepted and important contributor to BPD. Exposure to oxygen and positive pressure ventilation leads to developmental arrest and parenchymal injury in the immature preterm lung. Because even brief exposure to intubated positive pressure ventilation is injurious, avoiding invasive mechanical ventilation is the most widely acknowledged strategy to prevent VILI and the long-term sequela of BPD. Therefore, time on ventilators and rates of successful extubation are important endpoints of therapy.

Non-invasive neurally adjusted ventilatory assist (NIV-NAVA) is an FDA approved technology that consistently synchronizes non-invasive respiratory support with infant respiratory drive. The Diaphragmatic Initiated Ventilatory Assist (DIVA) trial is an unblinded, pragmatic, multicenter phase III randomized clinical trial in extremely preterm infants 23 0/7- 28 6/7 weeks gestational age to determine if NIV-NAVA, compared with non-synchronized nasal intermittent positive pressure ventilation (NS-NIPPV), prevents extubation failure within 5 days (120 hours) of extubation from mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 23 0/7- 28 6/7 weeks at birth
* Intubated in the first 7 days of life
* Undergoing extubation following at least 12 hours of invasive mechanical ventilation
* Post-natal age <32 weeks Post menstrual age at time of extubation

Exclusion Criteria:

* Major congenital anomalies, including pulmonary hypoplasia
* Neurologic disorders affecting respiratory drive (other than apnea of prematurity)
* Esophageal bleeding or other contraindication to NG/OG catheter placement
* Current weight <500 grams (based on Edi catheter approval)
* Study ventilator not available at time eligibility criteria are met
* Planned surgery or invasive procedure within 5 days of extubation
* Informed consent not provided

Ages: 0 Days to 9 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 478 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | within the first 5 days (120 hours) post extubation
  Extubation failure is defined when an infant is on the allocated mode of respiratory support and meets any of the following 4 criteria: (1) Rise in FiO2 at least 20% from pre-extubation value for >2 hours to maintain local SpO2 targets, (2) pH ≤7.20 or pCO2 ≥70mm Hg; (3) >1 apneic event requiring positive pressure ventilation (PPV) within 6 hours or ≥ 6 apneic events requiring stimulation within 6 hours (4) emergent intubation by the clinical team for cardiovascular instability or surgery.

SECONDARY OUTCOMES:
Bronchopulmonary Dysplasia (BPD) at 36 weeks PMA | 36 weeks PMA
  BPD will be assessed as an ordinal outcome (none, grade 1, 2, 3), according to the NRN criteria.
Death or BPD at 36 weeks PMA | 36 weeks PMA
  Composite dichotomous (y/n) outcome of death or grade 2/3 BPD, using the NRN criteria
Endotracheal intubation through 36 weeks PMA | 36 weeks PMA
  Endotracheal intubation will be assessed 2 ways: As a dichotomous (y/n) outcome if it occurs at any time and also as days until endotracheal intubation (with censoring at 36 weeks PMA)
Postmenstrual age at last invasive ventilation | 36 weeks PMA
  Time to cessation of invasive ventilation, with censoring at 36 weeks PMA
Postmenstrual age at last positive pressure support | 36 weeks PMA
  Time to cessation of positive pressure respiratory support, with censoring at 36 weeks PMA
Postmenstrual age at last supplemental oxygen | 36 weeks PMA
  Time to cessation of supplemental oxygen, with censoring at 36 weeks PMA
Prematurity-related morbidities through 36 weeks PMA | 36 weeks PMA
  Brain injury (intraventricular hemorrhage and periventricular leukomalacia), patent ductus arteriosus requiring therapy, pulmonary hemorrhage, culture proven sepsis, necrotizing enterocolitis, retinopathy of prematurity

OTHER OUTCOMES:
Death | From randomization through 36 weeks PMA
  Death will be measured in two ways (1) as a dichotomous (y/n) outcome if death occurs prior to 36 weeks PMA, and (2) days until death (with censoring at 36 weeks PMA).
Air Leaks | From randomization through 36 weeks PMA
  Air leaks will be measured as a dichotomous (y/n) outcome if a new pulmonary interstitial emphysema or pneumothorax occurs at any time after randomization until 36 weeks PMA.
Gastrointestinal perforation or bleeding | From randomization through 36 weeks PMA
  This will be measured as a dichotomous (y/n) outcome if a new GI perforation or bleeding occurs at any time after randomization until 36 weeks PMA.
Regional distribution of lung aeration | From extubation through 5 days after extubation
  this will be measured with electrical impedance tomography in a subset of patients
Mean airway pressure | From extubation through 5 days after extubation
  this will be measured from ventilator downloads for a subset of patients
peak inflation pressure | From extubation through 5 days after extubation
  this will be measured from ventilator downloads for a subset of patients
Edi signal | From extubation through 5 days after extubation
  this will be measured from ventilator downloads for a subset of patients
Fio2 | From extubation through 5 days after extubation
  this will be measured from ventilator downloads for a subset of patients

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Foglia, Principal Investigator — CHOP/UPENN
Locations (20):
- United States (17):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University, Loma Linda, California
  - Sharp Mary Birch, San Diego, California
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - AdventHealth, Orlando, Florida
  - Peyton Manning Children's Hospital, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University in St.Louis, St Louis, Missouri
  - Virtua Vorhees Hospital, Voorhees Township, New Jersey
  - Levine Children's Hospital, Charlotte, North Carolina
  - Atrial Health Brenner Children's Hospital( Wake Forest), Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Hospital, Provo, Utah
  - Children's Hospital of Richmond, Richmond, Virginia
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mt Sinai Hospital, Toronto
  - BC Children's and Women's Hospital, Vancouver

IPD SHARING:
Plan to Share IPD: Yes
Research records will be retained at each study site, and at the DCC for 3 years after completion of the study. We will follow NIH sharing policies with regards to sharing of data and specimens to public repositories, where appropriate
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years after completion of the study

REFERENCES:
- [Derived] Matlock DN, Ratcliffe SJ, Courtney SE, Kirpalani H, Firestone K, Stein H, Dysart K, Warren K, Goldstein MR, Lund KC, Natarajan A, Demissie E, Foglia EE. The Diaphragmatic Initiated Ventilatory Assist (DIVA) trial: study protocol for a randomized controlled trial comparing rates of extubation failure in extremely premature infants undergoing extubation to non-invasive neurally adjusted ventilatory assist versus non-synchronized nasal intermittent positive pressure ventilation. Trials. 2024 Mar 20;25(1):201. doi: 10.1186/s13063-024-08038-4. PMID 38509583